CLINICAL TRIAL: NCT02935907
Title: A Phase I Study of the Safety, Pharmacokinetic and Pharmacodynamic Properties of Orally Administered APG-115 in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: APG-115 in Patients With Advanced Solid Tumors or Lymphomas
Acronym: APG-115
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-115-US-001
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Patients With Advanced Solid Tumor or Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- APG-115 (Experimental): APG-115 to be explored sequentially during accelerated dose escalation. This will continue until either the occurrence in Cycle 1 of one DLT or two Grade 2 toxicities (graded as per the National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.0) that are related or possibly related to APG-115. When either of these criteria is fulfilled, dose escalation will be converted to a standard 3+3 escalation scheme,
  Interventions: Drug: APG-115

INTERVENTIONS:
Drug: APG-115 — Multiple dose cohorts, PO, every other day of a 28 day cycle

SUMMARY:
APG-115 is a novel, orally active small-molecule mouse double minute 2 homolog (MDM2) inhibitor. Mechanistically, APG-115 increases p53 and p21 overexpression, activates p53 - mediated apoptosis in tumor cells retaining wild-type p53. APG-115 has shown strong dose- and schedule-dependent antitumor activities in multiple human cancer xenograft and a patient derived xenograft (PDX) models. The preclinical data generated from APG-115 suggest that it may have a broad therapeutic potential for the treatment of human cancer as a single agent and in combination with other classes of anticancer drugs. APG-115 is intended for the treatment of patients with advanced solid tumors and lymphomas. Upon completion of the Phase 1 dose escalation study to establish the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and/or recommended phase 2 dose (RP2D), several phase Ib/II studies will be implemented accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic solid tumor or lymphoma that has relapsed from or is refractory to standard treatment, or no standard treatment is available. Only patients with advanced/metastatic cancer who have disease progression after treatment with all available therapies that are known to confer clinical benefit.
2. Male or non-pregnant, non-lactating female patients age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
4. Adequate hematologic and bone marrow functions
5. Adequate renal and liver function
6. Troponin (I) ≤ Upper Limit of Normal
7. Brain metastases with clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function & no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.
8. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug.
9. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
10. Willingness and ability to comply with study procedures and follow-up examination.
11. Willingness to provide and there is confirmed availability of pre-existing diagnostic or resected tumor samples, such as paraffin-embedded sections. Providing fresh tumor biopsy is optional for subjects in dose escalation cohorts.
12. Willingness to undergo tumor genotyping for P53 mutation at screening. Confirmation of P53 non-mutant status is encouraged, but not required.

Exclusion Criteria:

1. Receiving concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, with the exception of hormones for hypothyroidism or estrogen replacement therapy (ERT), anti estrogen analogs, agonists required to suppress serum testosterone levels); or any investigational therapy within 14 days prior to the first dose of study drug.
2. Steroid therapy for anti-neoplastic intent within 7 days prior to the first dose of study drug.
3. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to ≤ Grade 2.
4. Has gastrointestinal conditions that could affect the absorption of APG-115 in the opinion of the Investigator.
5. Use of therapeutic doses of anti-coagulants is excluded, along with anti-platelet agents; low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter are permitted.
6. Received a biologic (granulocyte colonystimulating factor, granulocyte-macrophage colony-stimulating factor or erythropoietin) within 14 days prior to the first dose of study drug.
7. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
8. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry.
9. Neurologic instability per clinical evaluation due to tumor involvement of the central nervous system (CNS). Patients with CNS tumors that have been treated, are asymptomatic and who have discontinued steroids (for the treatment of CNS tumors) for > 28 days may be enrolled.
10. Active symptomatic fungal, bacterial and/or viral infection including, but not limited to, active human immunodeficiency virus (HIV) or viral hepatitis (B or C).
11. Diagnosis of fever and neutropenia within 1 week prior to study drug administration.
12. Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
13. Prior treatment with MDM2 inhibitors.
14. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Patients with APG-115 treatment related adverse events (AE), serious adverse events (SAE) will be assessed according NCI CTCAE Version 4.0

SECONDARY OUTCOMES:
Response will be evaluated every 2 cycles (8 weeks), according to the revised RECIST Guideline, Version 1.1 | 18-24 months
Maximum plasma concentration (Cmax) of APG-115 on Day 1-3 and Day 21-23 post APG-115 treatment on cycle 1 | 23 days
Area under the plasma concentration versus time curve (AUC) of APG-115 on Day 1 -3 and Day 21 - 23 post APG-115 treatment on cycle 1 | 23 days

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (2):
- United States (2):
  - START Midwest, Grand Rapids, Michigan
  - The START Center for Cancer Care, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No